CLINICAL TRIAL: NCT03034018
Title: A Double-blind, Randomized, Placebo-controlled Study to Determine the Efficacy of Suvorexant in the Treatment of Hot Flash-associated Insomnia in Midlife Women
Brief Title: Efficacy of Suvorexant in the Treatment of Hot Flash-associated Insomnia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Hadine Joffe, MD MSc, Executive Director, Connors Center for Women's Health and Gender Biology, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016P002667
Record Dates: First submitted 2017-01-25; First posted 2017-01-27 (Estimated); Results first posted 2021-10-29 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Insomnia
Keywords: insomnia; hot flashes; menopause; suvorexant; belsomra
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Hot Flashes | interventions — suvorexant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- suvorexant (Experimental): suvorexant 10-20 mg taken at bedtime for four weeks
  Interventions: Drug: suvorexant
- placebo (Placebo Comparator): placebo taken at bedtime for four weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: suvorexant — 10-20 mg taken at bedtime for four weeks
  Other Names: Belsomra
  Arms: suvorexant
Drug: placebo — placebo taken at bedtime for four weeks
  Arms: placebo

SUMMARY:
The aim of this study is to determine the effect of suvorexant on insomnia symptoms in peri- and postmenopausal women who are experiencing sleep difficulties related to nighttime hot flashes.

ELIGIBILITY:
Inclusion Criteria:

* Peri- or postmenopausal women
* DSM-5 criteria for Insomnia disorder, with onset of symptoms attributed to hot flashes
* Some awakenings co-occur with a hot flash
* Score on the Insomnia Severity Index (ISI) measure ≥15
* Hot flashes present, including at night

Exclusion Criteria:

* Diagnosis of other primary sleep disorders
* Shift workers
* Current or expected use of hypnotic medications
* Current major depressive episode
* Lifetime history of bipolar disorder, psychosis, or other serious mental health problem
* Current alcohol/substance use disorder
* Obesity
* Renal or hepatic disease
* Pregnancy or breastfeeding
* Recent malignancy
* Recent surgery
* Neurological disorder or cardiovascular disease raising safety concerns
* Medical instability considered to interfere with study procedures
* Concomitant medications with drug interaction or co-administration concerns
* Contraindications or allergic responses to suvorexant
* Recent or planned travel across time zones
* Excessive coffee or cigarette use

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2020-04-03 (Actual); Study Completion 2020-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hadine Joffe, MD MSc, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Rahman SA, Nathan MD, Wiley A, Crawford S, Cohn AY, Harder JA, Grant LK, Erickson A, Srivastava A, McCormick K, Bertisch SM, Winkelman JW, Joffe H. A double-blind, randomized, placebo-controlled trial of suvorexant for the treatment of vasomotor symptom-associated insomnia disorder in midlife women. Sleep. 2022 Mar 14;45(3):zsac007. doi: 10.1093/sleep/zsac007. PMID 35022783

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Suvorexant | Placebo
Started | 30 | 30
Initiated Assigned Treatment | 27 | 29
Completed | 25 | 28
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Suvorexant | Placebo | Total
Number analyzed (Participants) | 27 | 29 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 29 | 56
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (4.5) | 53.4 (3.9) | 54.3 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 29 | 56
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 24 | 23 | 47
  Unknown or Not Reported | 2 | 4 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 4 | 4
  White | 25 | 20 | 45
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 4 | 5
Region of Enrollment [Number; unit: participants]
  United States | 27 | 29 | 56

OUTCOME MEASURES:

1. Primary Outcome: Within-person Change in ISI Score
Description: The Insomnia Severity Index (ISI) is a scale comprising seven questions scored 0-3. The total ISI score is the sum of all questions, with a total range from 0-21 with higher values indicating worse insomnia. Within-person change in ISI score from baseline to 4 weeks was calculated.
Time Frame: baseline and 4 weeks
Population: Participants who initiated treatment
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 27 | 29
score on a scale | -8.1 [-10.2 to -6.0] | -5.6 [-7.4 to -3.9]

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Suvorexant | Placebo
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/29
Other Adverse Events (participants affected / at risk) | 10/27 | 6/29
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Suvorexant (N=27) | Placebo (N=29)
somnolence (General disorders) | 4 (4) | 1 (1)
dry mouth (General disorders) | 3 (3) | 2 (2)
gastro-intestinal symptoms (Gastrointestinal disorders) | 2 (2) | 1 (1)
mood symptoms (Psychiatric disorders) | 2 (2) | 1 (1)
headache (General disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-09): https://cdn.clinicaltrials.gov/large-docs/18/NCT03034018/Prot_SAP_000.pdf